CLINICAL TRIAL: NCT02965599
Title: A Randomised, Multi-center, Double Blind (Sponsor Open), Placebo-controlled Study to Assess the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK3117391 in Subjects With Severe, Active Rheumatoid Arthritis
Brief Title: Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK3117391 in Subjects With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated following an internal review of the company's current research and development portfolio.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 204957; 2015-005800-27 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: pharmacodynamics; tolerability; GSK3117391; safety; efficacy; rheumatoid arthritis; pharmacokinetics
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK3117391 (Experimental): Subjects will receive GSK3117391 (Dose A) for 28 days.
  Interventions: Drug: GSK3117391
- Placebo (Placebo Comparator): Subjects will receive placebo for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3117391 — GSK3117391 (Dose A) is a white, opaque, gelatin capsule.
  Arms: GSK3117391
Drug: Placebo — Placebo is a white, opaque, gelatin capsule.
  Arms: Placebo

SUMMARY:
GSK3117391 has the potential to complement existing therapies in the treatment of chronic inflammatory disorders such as rheumatoid arthritis (RA). This study will evaluate the efficacy, safety and tolerability of oral GSK3117391 (Dose A) administered to subjects with severe RA despite treatment with disease-modifying anti-rheumatic drugs (DMARDs). This is a randomised, double-blind (sponsor open), multicentre, placebo-controlled, parallel group study. The total maximum study duration is approximately 10 weeks. Following a screening period of up to 28 days, subjects will be randomized (1:1) to placebo or GSK3117391 (Dose A) administered orally for a period of 28 days. Subjects will be followed up for 7 to 14 days post final dose. Approximately 40 subjects with severe RA will be randomised into the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years at the time of signing the informed consent.
* The subject must have a diagnosis of RA according to the 2010 ACR/ European League Against Rheumatism (EULAR) classification criteria for RA.
* Functional class I, II or III defined by the 1992 ACR Classification of Functional Status in RA
* The subject must have a EULAR DAS 28-CRP of greater than 5.1 at screening.
* Disease duration of >6 months (time from onset of patient-reported symptoms of either pain or stiffness or swelling in hands, feet or wrists).
* Swollen joint count of >=6 (66-joint count) and tender joint count of >=8 (68-joint count) at screening and at day 1
* The subject must have a CRP serum level of >=5 mg/L at screening
* The subject has had an inadequate response or intolerance of DMARDs (due to lack of efficacy or toxicity, after at least 8 weeks treatment).
* Body weight >=45 kilograms (kg) and body mass index (BMI) within the 18.5 - 35 kg/square metre (m^2) inclusive.
* Male or female requirements. Males: Male subjects with female partners of child bearing potential must comply with contraception requirements from the time of first dose of study medication 91 days after the last dose of study medication. In addition, male subjects must not donate sperm for 91 days after the last dose of study medication.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

* Non-reproductive potential defined as pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea.
* Females of reproductive potential must have proper and established use of a Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 28 days prior to the first dose of study medication and until 15 weeks after the last dose of study medication and completion of the follow-up visit. In addition, subjects will be required to utilise a barrier method of contraception. A negative HCG pregnancy test, (serum at screening visit and urine for subsequent visits) with a sensitivity of at least 25 international units per litre [IU/L]) is required at the screening visit, between Day -7 to -4 and on Day 1 prior to dose administration. Further pregnancy tests are required at the weekly study visits and the follow-up visit.

  * Capable of giving signed informed consent that includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Pregnant or lactating women.
* Subjects who meet diagnostic criteria for any other rheumatic disease (example [eg], lupus erythematosus, gout, psoriatic arthritis).
* Subjects who have previously been treated with more than 1 biologic agent (such as TNF inhibitors eg. adalimumab, etanercept, infliximab, certolizumab, golimumab or non-TNF inhibitors eg. abatacept, rituximab, tociluzimab) or any investigational biologic.
* Subjects with past history of granulomatous disease eg. leprosy, sarcoidosis.
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, haematological (including clotting disorders), gastrointestinal (including gastrooesophageal ulcers), pulmonary, cardiac (including ischemic heart disease), neurological, or cerebral disease, or other medical conditions that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study.
* Subjects with any values for monocytes are below the lower limit of normal (LLN) at screening.
* Haemoglobin <11 grams (g)/decilitre (dL); haematocrit <30%, white blood cell count <=3,000/cubic millimeter (mm^3) (<=3.0 x 10^9/litre [L]) or >=14,000/mm^3 (>=14 x 10^9/L); platelet count <= 100,000/microlitre (μL) (<=100x10^9/L); absolute neutrophil count <=2x10^9/L; lymphocyte count <1x10^9/L at screening.
* Alanine transaminase (ALT) and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) by Fridericia's correction formula (QTcF) or QTc by Bazett's correction formula (QTcB) >450 milliseconds (msec) (based on the average of triplicate electrocardiograms [ECGs]) at screening.
* Abnormal findings on ECG considered clinically significant by the investigator.
* A history of carcinoma in situ and malignant disease, except for adequately treated non-invasive cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency.
* Abnormal chest X-ray within 12 weeks of Day 1 (locally read and reported by a radiologist) judged by the investigator as clinically-significant.
* History of infected joint prosthesis at any time, with the prosthesis still in situ. History of leg ulcers, catheters, chronic sinusitis or recurrent chest or urinary tract infections.
* Active infections, or history of recurrent infections (excluding recurrent fungal infections of the nail bed), or have required management of acute or chronic infections as follows:

  * Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).
  * Hospitalisation for treatment of infection within 12 weeks of Day 1.
  * Use of parenteral (intravenous [IV] or intramuscular [IM]) antimicrobials (antibacterials, antivirals, antifungals, or antiparasitic agents) within 12 weeks of Day 1 or oral antimicrobials within 14 days of Day 1.
* Any surgical procedure, including bone or joint surgery/synovectomy within 12 weeks prior to Day 1 or any planned surgery within the duration of the study or follow-up period.
* A vaccination (live or attenuated) within 30 days of Day 1 or Bacillus Calmette-Guérin (BCG) vaccination within 365 days of Day 1, or a live vaccination planned during the course of the study.
* The subject has received treatment with the therapies prohibited or changes to those treatments in the prescribed timeframe. Subjects who have previously taken >1 biologic therapy for RA are excluded from this study.
* Other medications (including vitamins, herbal and dietary supplements) will be considered on a case-by-case basis, and will be allowed if in the opinion of the investigator the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 millilitre [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Smokers who would not be able to refrain from smoking whilst in the clinic.
* Subjects who cannot refrain from consuming any of the following fruits or juices (alone or in combination): seville oranges, grapefruit, pummelos, or any citrus fruits from 7 days prior to the first dose of study medication until their discharge from the unit after their last dose of study medication.
* History of sensitivity to any components of the study medication, or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Serologic evidence of current/previous Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg) and anti-Hepatitis B core (anti-HBc) antibody as follows within 6 weeks of Day 1: Subjects positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded
* Hepatitis C: Positive test for Hepatitis C virus (HCV) antibody confirmed on a subsequent blood sample by Ribonucleic acid (RNA)-polymerase chain reaction (PCR) assay within 6 weeks of Day 1. Subjects who are positive for Hepatitis C antibody and negative for Hepatitis C RNA-PCR assay performed on a subsequent sample will be eligible to participate. Subjects who are positive for Hepatitis C antibody and have a positive result for Hepatitis C RNA-PCR assay performed on the subsequent sample,will not be eligible to participate.
* A positive test for HIV 1 or 2 at screening.
* Evidence of active or latent infection with Mycobacterium tuberculosis (TB), as defined by all of the following:

  * No history of active or latent TB infection irrespective of treatment status
  * A negative diagnostic TB test within 28 days of baseline (Day 1) defined as: A negative QuantiFERON Gold test or T-spot test (two successive indeterminate QuantiFERON tests will be considered as a positive result) OR If QuantiFERON gold or T-spot test not approved or registered in country of participation, then a negative tuberculin skin test (TST) reaction as per local guidelines is required (it is strongly recommended that subjects with a history of BCG vaccination be tested with QuantiFERON gold test).
  * Chest X-ray within 12 weeks of Day 1 with no evidence of current or previous pulmonary tuberculosis, locally read by a radiologist.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Participation in a trial with any investigational drug within 3 months or 5 half-lives (whichever is longer) before the start of the study and within 4 months if the study drug was new chemical entity. Exposure to more than 3 new chemical entities in a clinical study setting within 12 months prior to the first dosing day.
* Donation of blood in excess of 500 mL within a 56 day period prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Świdnik
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Târgu Mureş, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in participants with severe, active rheumatoid arthritis receiving GSK3117391, 40 milligrams (mg) or placebo at one center in Poland and one in Romania.
Pre-assignment Details: This study was terminated early by the sponsor following internal review. A total number of 26 participants were screened, of which three participants were enrolled in the study.
Groups:
- Placebo: Eligible participants in this arm, received a matching placebo to the study drug GSK3117391, administered orally once a day as 2 capsules in the morning, following every other day, for 28-days.
- GSK3117391, 40 mg: Eligible participants in this arm, received a dose of 40 mg of GSK3117391, administered orally once a day as 2 capsules of 20 mg each in the morning, following every other day, for 28-days.
Period: Overall Study
Arm/Group | Placebo | GSK3117391, 40 mg
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Protocol-defined stop criteria reached | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3117391, 40 mg | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (14.85) | 46 (NA) — NA indicates that SD could not be calculated for a single participant. | 54.3 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score for 28 Different Joints With (DAS28) C-reactive Protein (CRP) at Day 28
Description: The DAS28 score is a derived measurement with differential weighing given to each component as: Tender/Painful Joint Count (TJC28) and swollen joint count (SJC28) both scored 0-28 (higher scores indicate higher disease activity), CRP measured in milligrams per liter and Patient's Global Assessment of Arthritis (PtGA) (visual analogue scale with values from 0 [best] to 100 [worst]). The formula used to calculate DAS28 score was 0.56 multiplied by square root of TJC28 plus 0.28 multiplied by square root of SJC28 plus 0.36 log of (CRP plus 1) plus 0.014 multiplied by PtGA plus 0.96. DAS28 scores ranged from 0 (best) to 10 (worst). A negative change from Baseline value indicated improvement. Baseline was defined at Day 1 (pre-dose). Change from Baseline was post-baseline value minus the value at Baseline. Safety Population consisted of all participants who received at least one dose of study medication. Individual participant data at Day 28 has been presented.
Time Frame: Baseline (pre-dose, Day 1) and Day 28
Population: Safety Population. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Units on a scale
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 1 | 1
Units on a scale | -0.38 | -1.73

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect and other situations which involve medical or scientific judgment, and is associated with liver injury and impaired liver function.
Time Frame: Up to Day 44
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Participants
  Any non-SAE | 2 | 0
  Any SAE | 0 | 0

3. Secondary Outcome: Number of Participants With Vital Signs Values of Potential Clinical Importance (PCI)
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP), temperature and heart rate were measured in semi-supine position after 5 minutes rest. The PCI ranges for vitals were as follows; for SBP <85 or >160 millimeters of mercury (mmHg), for DBP <45 or >100 mmHg, for heart rate <40 or >110 beats per minute and for temperature <36 or >38 Celsius. The number of participants with vital signs of PCI have been presented.
Time Frame: Up to Day 44
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Participants
  SBP | 0 | 0
  DBP | 0 | 0
  Heart rate | 0 | 0
  Temperature | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were performed during the study using an automated ECG machine, after 5 minutes of rest. The number of participants with abnormal ECG findings were reported and categorized as clinically significant and not clinically significant. Any value for ECG parameters out of the following normal range was considered as clinically significant abnormality; for PR interval <110 or >220 milliseconds, for QRS interval <75 or >110 milliseconds and for QT corrected interval <450 milliseconds.
Time Frame: Up to Day 44
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Participants
  Abnormal-clinically significant | 0 | 0
  Abnormal-Not clinically significant | 1 | 0

5. Secondary Outcome: Number of Participants With Values for Clinical Chemistry Parameters of PCI
Description: Blood samples were collected for analysis of clinical chemistry parameters. The PCI ranges were for Albumin <30 millimoles/Liter (mmol/L), Calcium (<2 or >2.75 mmol/L), Creatinine (>44.2 mmol/L), Glucose (<3 or >9 mmol/L), Magnesium (<0.5 or >1.23 mmol/L), Phosphorus (<0.8 or > 1.6 mmol/L), Potassium (<3 or > 5.5 mmol/L), Sodium (<130 or 150 mmol/L), Total carbon-dioxide (<18 or > 32 mmol/L), Alanine aminotransferase (>= 2x Upper Limit of Normal [ULN]), Aspartate aminotransferase (>=2x ULN), alkaline phosphatase (>=2x ULN), and total bilirubin (>=1.5xULN). The number of participants with values for clinical chemistry parameters of PCI have been presented
Time Frame: Up to Day 44
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Values for Hematology Parameters of PCI
Description: Blood samples were collected for analysis of hematology parameters. PCI ranges were for platelets (< 50 or >550 × 10^9 cells/L), white blood cell count (<3 or >14 × 10^9 cells/L), hemoglobin (<90 or >180 g/L), hematocrit (if proportion of red blood cells in blood was <0.3 or >0.54), lymphocytes (<0.5 × 10^9 cells/L), neutrophils (<1.0 × 10^9 cells/L) and monocytes (<0.2 or 1.5 × 10^9 cells/L). The number of participants with values for hematology parameters of PCI have been presented.
Time Frame: Up to Day 44
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Participants | 1 | 1

7. Secondary Outcome: Number of Participants With Abnormal Findings for Urinalysis Parameters
Description: Urine samples were collected for the analysis of specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones at specified time points. The number of participants with abnormal urinalysis findings have been presented.
Time Frame: Up to Day 44
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Criteria
Description: A participant was considered to be a responder according to the ACR20 criteria if the participant had at least 20% improvement in both the tender joint count and swollen joint count measures, and 20% improvement in at least 3 of the following 5 measures: patient and physician global assessments, pain, disability, and an acute-phase reactant. This analysis was planned but data was not collected , as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: Up to Day 44
Population: Safety Population. Data was not collected, as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants Achieving ACR 50, Criteria
Description: A participant was considered to be a responder according to the ACR50 criteria if the participant had at least 50% improvement in both the tender joint count and swollen joint count measures, and 50% improvement in at least 3 of the following 5 measures: patient and physician global assessments, pain, disability, and an acute-phase reactant. This analysis was planned but data was not collected , as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: Up to Day 44
Population: as for outcome 8
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants Achieving ACR 70, Criteria
Description: A participant was considered to be a responder according to the ACR70 criteria if the participant had at least 70% improvement in both the tender joint count and swollen joint count measures, and 70% improvement in at least 3 of the following 5 measures: patient and physician global assessments, pain, disability, and an acute-phase reactant. This analysis was planned but data was not collected , as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: Up to Day 44
Population: as for outcome 8
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Swollen Joints Assessed Using 28-joint Counts
Description: The total number of joints ranging from 0 to 28 joints with a present swelling were assessed. The following 28 joints were taken into account for SJC28: Shoulder (2 joints), Knee (2), Elbow (2), Wrist (2), Fingers (Joints for proximal interphalangeal [PIP] and metacarpophalangeal [MCP]: 20). No missing observations were considered. Individual participant data has been presented. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Days 1, 7, 14, 21, 28 and Follow-up (Day 44)
Population: Safety Population. Only those participants with data available at specified time point has been analyzed (represented by n=x in category titles). Data has been presented for participants as per the actual treatment received.
Measure: Number; unit: Swollen joints
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Swollen joints
  Participant 1; Day 1; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 1; n=1,0 | 7 |
  Participant 1; Day 7; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 7; n=1,0 | 2 |
  Participant 1; Follow-up (Day 44); n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Follow-up (Day 44); n=1,0 | 1 |
  Participant 2; Day 1; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 1; n=1,0 | 8 |
  Participant 2; Day 7; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 7; n=1,0 | 7 |
  Participant 2; Day 14; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 14; n=1,0 | 4 |
  Participant 2; Day 21; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 21; n=1,0 | 1 |
  Participant 2; Day 28; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 28; n=1,0 | 1 |
  Participant 2; Follow-up (Day 44); n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Follow-up (Day 44); n=1,0 | 1 |
  Participant 3; Day 1;n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 1;n=0,1 |  | 28
  Participant 3; Day 7;n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 7;n=0,1 |  | 18
  Participant 3; Day 14;n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 14;n=0,1 |  | 12
  Participant 3; Day 21;n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 21;n=0,1 |  | 7
  Participant 3; Day 28;n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 28;n=0,1 |  | 11
  Participant 3; Follow-up (Day 44);n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Follow-up (Day 44);n=0,1 |  | 5

12. Secondary Outcome: Number of Tender/Painful Joints Assessed Using 28-joint Counts
Description: The total number of joints ranging from 0 to 28 joints with a present tenderness were assessed. The following 28 joints were taken into account for TJC28: Shoulder (2 joints), Knee (2), Elbow (2), Wrist (2), Fingers (PIP and MCP: 20). No missing observations were considered. Individual participant data has been presented. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Days 1, 7, 14, 21, 28 and Follow-up (Day 44)
Population: as for outcome 11
Measure: Number; unit: Tender/painful joints
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Tender/painful joints
  Participant 1; Day 1; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 1; n=1, 0 | 12 |
  Participant 1; Day 7; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 7; n=1, 0 | 8 |
  Participant 1; Follow-up (Day 44); n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Follow-up (Day 44); n=1, 0 | 1 |
  Participant 2; Day 1; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 1; n=1, 0 | 9 |
  Participant 2; Day 7; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 7; n=1, 0 | 7 |
  Participant 2; Day 14; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 14; n=1, 0 | 5 |
  Participant 2; Day 21; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 21; n=1, 0 | 7 |
  Participant 2; Day 28; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 28; n=1, 0 | 4 |
  Participant 2; Follow-up (Day 44); n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Follow-up (Day 44); n=1, 0 | 1 |
  Participant 3; Day 1; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 1; n=0,1 |  | 28
  Participant 3; Day 7; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 7; n=0,1 |  | 26
  Participant 3; Day 14; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 14; n=0,1 |  | 19
  Participant 3; Day 21; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 21; n=0,1 |  | 18
  Participant 3; Day 28; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 28; n=0,1 |  | 19
  Participant 3; Follow-up (Day 44); n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Follow-up (Day 44); n=0,1 |  | 8

13. Secondary Outcome: Change From Baseline in DAS28-CRP Over Time
Description: The DAS28 score is a derived measurement with differential weighing given to each component as: TJC28 and SJC28 both scored 0-28 (higher scores indicate higher disease activity), CRP measured in milligrams per liter and PtGA (visual analogue scale with values from 0 [best] to 100 [worst]). The formula used to calculate DAS28 score was 0.56 multiplied by square root of TJC28 plus 0.28 multiplied by square root of SJC28 plus 0.36 log of (CRP plus 1) plus 0.014 multiplied by PtGA plus 0.96. DAS28 scores ranged from 0 (best) to 10 (worst). A negative change from Baseline value indicated improvement. Baseline was defined at Day 1 (pre-dose). Change from Baseline was post-baseline value minus the value at Baseline. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Baseline (pre-dose, Day 1) and Days 7, 14, 21, 28, Follow-up (Day 44)
Population: as for outcome 11
Measure: Number; unit: Scores on a Scale
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Scores on a Scale
  Participant 1; Day 7 ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 7 ;n=1, 0 | -0.48 |
  Participant 1; Follow-up (Day 44) ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Follow-up (Day 44) ;n=1, 0 | -2.84 |
  Participant 2; Day 7 ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 7 ;n=1, 0 | -0.24 |
  Participant 2; Day 14 ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 14 ;n=1, 0 | -0.96 |
  Participant 2; Day 21 ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 21 ;n=1, 0 | -0.77 |
  Participant 2; Day 28 ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 28 ;n=1, 0 | -0.38 |
  Participant 2; Follow-up (Day 44) ;n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Follow-up (Day 44) ;n=1, 0 | -2.30 |
  Participant 3; Day 7 ;n=0, 1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 7 ;n=0, 1 |  | -0.79
  Participant 3; Day 14 ;n=0, 1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 14 ;n=0, 1 |  | -1.35
  Participant 3; Day 21 ;n=0, 1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 21 ;n=0, 1 |  | -1.54
  Participant 3; Day 28 ;n=0, 1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 28 ;n=0, 1 |  | -1.73
  Participant 3; Follow-up (Day 44) ;n=0, 1: number analyzed (Participants) | 0 | 1
  Participant 3; Follow-up (Day 44) ;n=0, 1 |  | -2.59

14. Secondary Outcome: Assessment of Disease Activity Using Patient's Global Assessment of Arthritis (PtGA)
Description: Participants completed the global assessment of disease activity using the PtGA item using visual analogue scale (VAS) ranging from "0" (none) to "100" (extremely active), respectively. Individual participant score has been presented. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Days 1, 7, 14, 21, 28 and Follow-up (Day 44)
Population: as for outcome 11
Measure: Number; unit: Scores on a Scale
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Scores on a Scale
  Participant 1; Day 1; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 1; n=1, 0 | 58 |
  Participant 1; Day 7; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 7; n=1, 0 | 73 |
  Participant 1; Follow-up (Day 44); n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Follow-up (Day 44); n=1, 0 | 25 |
  Participant 2; Day 1; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 1; n=1, 0 | 87 |
  Participant 2; Day 7; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 7; n=1, 0 | 86 |
  Participant 2; Day 14; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 14; n=1, 0 | 71 |
  Participant 2; Day 21; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 21; n=1, 0 | 78 |
  Participant 2; Day 28; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 28; n=1, 0 | 96 |
  Participant 2; Follow-up (Day 44); n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Follow-up (Day 44); n=1, 0 | 33 |
  Participant 3; Day 1; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 1; n=0,1 |  | 100
  Participant 3; Day 7; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 7; n=0,1 |  | 82
  Participant 3; Day 14; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 14; n=0,1 |  | 79
  Participant 3; Day 21; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 21; n=0,1 |  | 74
  Participant 3; Day 28; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 28; n=0,1 |  | 72
  Participant 3; Follow-up (Day 44); n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Follow-up (Day 44); n=0,1 |  | 62

15. Secondary Outcome: Change From Baseline in CRP
Description: Blood samples were collected at indicated time points for the analysis of CRP. Change from Baseline, was defined as the post-baseline value minus the value at Baseline. Baseline was defined as the value from the Day 1 (pre-dose). Individual participant data has been presented. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Baseline (pre-dose, Day 1) and Days 7, 14, 21, 28, Follow-up (Day 44)
Population: as for outcome 11
Measure: Number; unit: Milligrams per liter
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Milligrams per liter
  Participant 1; Day 7; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 7; n=1, 0 | 0.50 |
  Participant 1; Follow-up (Day 44); n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 1; Follow-up (Day 44); n=1, 0 | -11.20 |
  Participant 2; Day 7; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 7; n=1, 0 | 0.50 |
  Participant 2; Day 14; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 14; n=1, 0 | -1.60 |
  Participant 2; Day 21; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 21; n=1, 0 | 1.60 |
  Participant 2; Day 28; n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 28; n=1, 0 | 30.20 |
  Participant 2; Follow-up (Day 44); n=1, 0: number analyzed (Participants) | 1 | 0
  Participant 2; Follow-up (Day 44); n=1, 0 | 2.20 |
  Participant 3; Day 7; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 7; n=0,1 |  | -14.00
  Participant 3; Day 14; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 14; n=0,1 |  | -3.10
  Participant 3; Day 21; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 21; n=0,1 |  | 23.40
  Participant 3; Day 28; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 28; n=0,1 |  | -22.40
  Participant 3; Follow-up (Day 44); n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Follow-up (Day 44); n=0,1 |  | 26.70

16. Secondary Outcome: Plasma Concentrations of GSK3117391 and GSK3339189
Description: Blood samples were planned to be collected for GSK3117391 and its acid metabolite GSK3339189, at the specified timepoints. The Pharmacokinetic (PK) Population was defined as participants in the Safety Population who received an active dose and for whom a PK sample was obtained and analyzed. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 10 hours (Day 1) and 24 hours (Day 2) post-dose; pre-dose, 0.25, 0.5, 1, 4, and 8 hours (Day 3) post-dose; pre-dose (Day 7); pre-dose (Day 21); pre-dose, 0.25, 0.5, 1, 2, 4, 6, 10 hours (Day 27) and 24 hours post-dose
Population: PK Population. Data was not collected, as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Groups:
- GSK3339189: GSK3339189 is a metabolite of GSK3117391. Eligible participants in this arm, received a dose of 40 mg of GSK3117391, administered orally once a day as 2 capsules of 20 mg each in the morning, following every other day, for 28-days.
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Maximum Observed Blood Concentration (Cmax) of GSK3117391 and GSK3339189
Description: Cmax was defined as the maximum concentration of drug in the plasma. Blood samples were planned to be collected for GSK3117391 and its acid metabolite GSK3339189, at the specified time points. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Time to Cmax (Tmax)of GSK3117391 and GSK3339189
Description: Tmax was defined as time required to achieve Cmax for drug, in the plasma. Blood samples were planned to be collected for GSK3117391 and its acid metabolite GSK3339189, at the specified timepoints. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 10 hours (Day 1) and 24 hours (Day 2) post-dose; pre-dose, 0.25, 0.5, 1, 4, and 8 hours (Day 3) post-dose; pre-dose (Day 7); pre-dose (Day 21); pre-dose, 0.25 hour, 0.5, 1, 2, 4, 6, 10 hours (Day 27) and 24 hours post-dose
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC[0-t]) of GSK3117391 and GSK3339189
Description: Blood samples were planned to be collected for GSK3117391, and its acid metabolite GSK3339189, at the specified time points. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: as for outcome 18
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: AUC From Time Zero to the Time of Next Dosing (AUC[0- Tau]) of GSK3117391 and GSK3339189
Description: Blood samples were planned to be collected for GSK3117391 and its acid metabolite GSK3339189, at the specified timepoints. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: AUC From Time Zero to Infinity (AUC[0-infinity]) of GSK3117391 and GSK3339189
Description: as for outcome 20
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) of GSK3117391 and GSK3339189
Description: as for outcome 20
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Trough Concentration (Ctau) of GSK3117391 and GSK3339189
Description: as for outcome 20
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Observed Accumulation Ratio (Ro) of GSK3117391 and GSK3339189
Description: Blood samples were planned to be collected for GSK3117391, and its acid metabolite GSK3339189, at the specified timepoints. Accumulation ratio was planned to be determined from the ratio of AUC from time zero to time of next dosing (AUC [0-tau]) following single dose administration /AUC (0-tau) on repeat dose administration. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Apparent Total Clearance (CL/F) of GSK3117391 and GSK3339189
Description: CL/F, describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). Blood samples, were planned to be collected for GSK3117391, and its acid metabolite GSK3339189, at the specified timepoints. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Apparent Volume of Distribution (V/F) of GSK3117391 and GSK3339189
Description: V/F, is defined as the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma. Blood samples, were planned to be collected for GSK3117391, at the specified timepoints. This analysis was planned but was not performed as the sample size was too small and study was terminated pre-maturely, by the sponsor following internal review.
Time Frame: as for outcome 16
Population: as for outcome 16
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change From Baseline in Monocyte Count
Description: Blood samples were collected at the indicated time points for the analysis of monocytes. Change from Baseline was defined as the post-Baseline value minus the value at Baseline. Baseline was defined as the value from the Day 1 (pre-dose). Individual participant data has been presented. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Baseline (pre-dose, Day 1); 1, 4, 6, 10 Hours on Day 1; Day 2 (24 Hours); Pre-dose, 1, 4, 8 Hours on Day 3; Pre-dose on Day 7; Day 14; Pre-dose on Day 21; Pre-dose, 1, 4, 6, 10 Hours on Day 27; Day 28 (24 Hours); Day 30 (72 Hours) and Day 44 (Follow-up)
Population: as for outcome 11
Measure: Number; unit: Giga cells per liter
Arm/Group | GSK3339189 | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Giga cells per liter
  Participant 1; Day 1; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 1; 1 Hour; n=1,0 | -0.11 |
  Participant 1;Day 1; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 1; 4 Hours; n=1,0 | -0.04 |
  Participant 1;Day 1; 6 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 1; 6 Hours; n=1,0 | -0.34 |
  Participant 1;Day 1; 10 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 1; 10 Hours; n=1,0 | -0.13 |
  Participant 1;Day 3; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 3; Pre-dose; n=1,0 | -0.68 |
  Participant 1;Day 3; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 3; 1 Hour; n=1,0 | -0.59 |
  Participant 1; Day 3; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 3; 4 Hours; n=1,0 | -0.56 |
  Participant 1; Day 3; 8 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 3; 8 Hours; n=1,0 | -0.02 |
  Participant 1;Day 7; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 7; Pre-dose; n=1,0 | -0.25 |
  Participant 1;Follow-up (Day 44); n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Follow-up (Day 44); n=1,0 | 0.10 |
  Participant 2; Day 1; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 1; 1 Hour; n=1,0 | 0.25 |
  Participant 2;Day 1; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 1; 4 Hours; n=1,0 | 0.27 |
  Participant 2;Day 1; 6 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 1; 6 Hours; n=1,0 | 0.24 |
  Participant 2;Day 1; 10 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 1; 10 Hours; n=1,0 | 0.31 |
  Participant 2;Day 2; 24 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 2; 24 Hours; n=1,0 | 0.05 |
  Participant 2;Day 3; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 3; Pre-dose; n=1,0 | 0.27 |
  Participant 2;Day 3; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 3; 1 Hour; n=1,0 | 0.27 |
  Participant 2; Day 3; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 3; 4 Hours; n=1,0 | 0.24 |
  Participant 2; Day 3; 8 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 3; 8 Hours; n=1,0 | 0.05 |
  Participant 2;Day 7; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 7; Pre-dose; n=1,0 | 0.23 |
  Participant 2;Day 14; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 14; n=1,0 | 0.02 |
  Participant 2;Day 21; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 21; Pre-dose; n=1,0 | 0.12 |
  Participant 2;Day 27; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 27; Pre-dose; n=1,0 | 0.02 |
  Participant 2;Day 27; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 27; 1 Hour; n=1,0 | 0.23 |
  Participant 2;Day 27; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 27; 4 Hours; n=1,0 | 0.02 |
  Participant 2;Day 27; 6 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 27; 6 Hours; n=1,0 | -0.28 |
  Participant 2;Day 27; 10 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 27; 10 Hours; n=1,0 | 0.28 |
  Participant 2;Day 28; 24 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 28; 24 Hours; n=1,0 | 0.30 |
  Participant 2; Day 30; 72 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 30; 72 Hours; n=1,0 | 0.02 |
  Participant 2; Follow-up (Day 44); n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Follow-up (Day 44); n=1,0 | 0.09 |
  Participant 3; Day 1; 1 Hour; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 1; 1 Hour; n=0,1 |  | -0.84
  Participant 3;Day 1; 4 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 1; 4 Hours; n=0,1 |  | -0.14
  Participant 3;Day 1; 6 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 1; 6 Hours; n=0,1 |  | 0.29
  Participant 3;Day 1; 10 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 1; 10 Hours; n=0,1 |  | 0.30
  Participant 3;Day 2; 24 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 2; 24 Hours; n=0,1 |  | 0.29
  Participant 3;Day 3; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 3; Pre-dose; n=0,1 |  | -0.96
  Participant 3;Day 3; 1 Hour; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 3; 1 Hour; n=0,1 |  | -0.77
  Participant 3; Day 3; 8 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 3; 8 Hours; n=0,1 |  | -0.90
  Participant 3;Day 7; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 7; Pre-dose; n=0,1 |  | -0.79
  Participant 3;Day 14; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 14; n=0,1 |  | -1.11
  Participant 3;Day 21; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 21; Pre-dose; n=0,1 |  | -0.91
  Participant 3;Day 27; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 27; Pre-dose; n=0,1 |  | 0.10
  Participant 3;Day 27; 1 Hour; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 27; 1 Hour; n=0,1 |  | -0.99
  Participant 3;Day 27; 4 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 27; 4 Hours; n=0,1 |  | -0.97
  Participant 3;Day 27; 6 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 27; 6 Hours; n=0,1 |  | -0.14
  Participant 3;Day 27; 10 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 27; 10 Hours; n=0,1 |  | -1.06
  Participant 3;Day 28; 24 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 28; 24 Hours; n=0,1 |  | -0.94
  Participant 3; Day 30; 72 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 30; 72 Hours; n=0,1 |  | -0.91
  Participant 3; Follow-up (Day 44); n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Follow-up (Day 44); n=0,1 |  | -0.70

28. Secondary Outcome: Changes From Baseline in Soluble Cytokine
Description: Change from Baseline, was defined as the post-Baseline value minus the value at Baseline. Baseline was defined as the value from the Day 1 (pre-dose). Blood samples were planned to be analyzed by flow cytometry for cell markers to determine any changes after treatment with GSK3117391. This analysis was planned but the assay was not performed due to sample size being too small at the time of early study termination.
Time Frame: Baseline (pre-dose, Day 1) and up to 44 Days
Population: Safety Population. Data was not collected, assay was not performed due to sample size being too small at the time of early study termination.
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Changes From Baseline in Myeloid-related Protein 8/14 (MRP8/14)
Description: Blood samples were collected at the indicated time points and analyzed by flow cytometry for cell markers to determine any changes after treatment with GSK3117391. Change from Baseline was defined as the post-Baseline value minus the value at Baseline. Baseline was defined as the value from the Day 1 (pre-dose). Individual participant data has been presented. Only data available at specified visit with respect to the participant has been presented.
Time Frame: Baseline (pre-dose, Day 1); 1, 4, 10 Hours on Day 1; Day 2 (24 Hours); Pre-dose, 8 Hours on Day 3; Pre-dose on Day 7; Day 14; Pre-dose on Day 21; Pre-dose on Day 27; Day 28 (24 Hours) and Day 44 (Follow-up)
Population: as for outcome 11
Measure: Number; unit: Milligram per liter
Arm/Group | Placebo | GSK3117391, 40 mg
Number analyzed (Participants) | 2 | 1
Milligram per liter
  Participant 1; Day 1; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 1; 1 Hour; n=1,0 | -0.36 |
  Participant 1;Day 1; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 1; 4 Hours; n=1,0 | -0.57 |
  Participant 1;Day 1; 10 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 1; 10 Hours; n=1,0 | -0.46 |
  Participant 1;Day 2; 24 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 2; 24 Hours; n=1,0 | -0.52 |
  Participant 1;Day 3; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 3; Pre-dose; n=1,0 | -0.21 |
  Participant 1; Day 3; 8 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Day 3; 8 Hours; n=1,0 | -0.21 |
  Participant 1;Day 7; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1;Day 7; Pre-dose; n=1,0 | -0.39 |
  Participant 1; Follow-up (Day 44); n=1,0: number analyzed (Participants) | 1 | 0
  Participant 1; Follow-up (Day 44); n=1,0 | -1.22 |
  Participant 2; Day 1; 1 Hour; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 1; 1 Hour; n=1,0 | 0.27 |
  Participant 2;Day 1; 4 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 1; 4 Hours; n=1,0 | -1.13 |
  Participant 2;Day 1; 10 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 1; 10 Hours; n=1,0 | 0.37 |
  Participant 2;Day 2; 24 Hours;n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 2; 24 Hours;n=1,0 | -2.34 |
  Participant 2;Day 3; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 3; Pre-dose; n=1,0 | 0.20 |
  Participant 2; Day 3; 8 Hours;n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2; Day 3; 8 Hours;n=1,0 | -0.31 |
  Participant 2;Day 7; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 7; Pre-dose; n=1,0 | 2.29 |
  Participant 2;Day 14;n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 14;n=1,0 | 3.76 |
  Participant 2;Day 21; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 21; Pre-dose; n=1,0 | -0.78 |
  Participant 2;Day 27; Pre-dose; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 27; Pre-dose; n=1,0 | 0.67 |
  Participant 2;Day 28; 24 Hours; n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Day 28; 24 Hours; n=1,0 | -2.51 |
  Participant 2;Follow-up (Day 44); n=1,0: number analyzed (Participants) | 1 | 0
  Participant 2;Follow-up (Day 44); n=1,0 | -1.43 |
  Participant 3; Day 1; 1 Hour; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 1; 1 Hour; n=0,1 |  | -0.53
  Participant 3;Day 1; 4 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 1; 4 Hours; n=0,1 |  | 0.32
  Participant 3;Day 1; 10 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 1; 10 Hours; n=0,1 |  | 0.89
  Participant 3;Day 2; 24 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 2; 24 Hours; n=0,1 |  | 0.64
  Participant 3;Day 3; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 3; Pre-dose; n=0,1 |  | 2.95
  Participant 3; Day 3; 8 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3; Day 3; 8 Hours; n=0,1 |  | 7.06
  Participant 3;Day 7; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 7; Pre-dose; n=0,1 |  | 5.21
  Participant 3;Day 14; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 14; n=0,1 |  | 4.14
  Participant 3;Day 21; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 21; Pre-dose; n=0,1 |  | 5.90
  Participant 3;Day 27; Pre-dose; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 27; Pre-dose; n=0,1 |  | 1.41
  Participant 3;Day 28; 24 Hours; n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Day 28; 24 Hours; n=0,1 |  | -1.85
  Participant 3;Follow-up (Day 44); n=0,1: number analyzed (Participants) | 0 | 1
  Participant 3;Follow-up (Day 44); n=0,1 |  | -0.71

ADVERSE EVENTS:
Time Frame: All non-SAEs and SAEs were collected from start of the study treatment (Day 1) up to Day 44.
Description: The Safety Population was used to assess the non-SAEs and SAEs.
Arm/Group | Placebo | GSK3117391, 40 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | GSK3117391, 40 mg (N=1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT02965599/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT02965599/SAP_001.pdf